CLINICAL TRIAL: NCT01149109
Title: Phase III Trial of CCNU/Temozolomide (TMZ) Combination Therapy vs. Standard TMZ Therapy for Newly Diagnosed MGMT-methylated Glioblastoma Patients
Brief Title: Efficacy and Safety Study of Lomustine/Temozolomide Combination Therapy vs. Standard Therapy for Glioblastoma Patients
Acronym: CeTeG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Ulrich Herrlinger, Head, Division of Clinical Neurooncology, University Hospital, Bonn
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CeTeG; 2009-011252-22 (EudraCT Number)
Record Dates: First submitted 2010-06-14; First posted 2010-06-23 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Glioblastoma
Keywords: MGMT promotor status; overall survival
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide; Lomustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- lomustine (CCNU) + temozolomide (TMZ) and radiotherapy (Experimental): 60 Gy standard radiotherapy (RT, 30 x 2 Gy) Six 42-day courses of oral CCNU 100 mg/m2 (day 1) and oral TMZ 100 mg/m2 (day 2-6), first CCNU application during the first week of RT CCNU/TMZ and radiotherapy start 2-5 weeks after diagnosis (day of surgery for glioblastoma (GBM)). In courses 2-6, TMZ dose are adjusted according to the hematotoxicity observed in the previous course and can be increased stepwise up to 200 mg/m2/day
  Interventions: Drug: Temozolomide and lomustine
- temozolomide and radiotherapy (Active Comparator): 60 Gy standard radiotherapy (RT, 30 x 2 Gy) and concomitant TMZ therapy (daily TMZ 75 mg/m2) starting with the first day of radiotherapy Six 28-day courses of TMZ (day 1-5) starting 4 weeks after completion of radiotherapy. In the first course TMZ is given at a dose of 150 mg/m2/day, in case no toxicity is observed, the 2nd course is applied at a daily dose of 200 mg/m2
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: Temozolomide and lomustine
  Other Names: Temodal, Temomedac, CeCeNu
  Arms: lomustine (CCNU) + temozolomide (TMZ) and radiotherapy
Drug: Temozolomide
  Other Names: Temodal, Temomedac
  Arms: temozolomide and radiotherapy

SUMMARY:
The prognosis of patients with newly diagnosed glioblastoma is dismal despite recent therapeutic improvements Using standard therapy with temozolomide (TMZ) and radiotherapy (60 Gy), the median overall survival time (mOS) is 14.6 months (Stupp et al., 2005). Since in a previous non-randomized bicentric phase II trial, primary combination chemotherapy with lomustine (CCNU) and TMZ was highly effective (mOS 23 months; UKT-03 trial; Herrlinger et al., 2006; Glas et al., 2009) the proposed trial further investigates the efficacy of CCNU/TMZ in a randomized multicenter phase III setting against standard therapy. In case the projected phase III trial confirms the phase II data, CCNU/TMZ combination would be significantly better than TMZ monotherapy and would thus be the new standard treatment for newly diagnosed GBM patients with a methylated MGMT promotor. Thus, this trial has the potential to profoundly change the standard therapy of this most aggressive brain tumor. Since in the previous trial only patients with a methylated MGMT (mMGMT) promoter had a benefit from CCNU/TMZ (mOS in the mMGMT group 34 months, in the non-mMGMT group 12.5 months; Glas et al., 2009) while patients with a non-methylated MGMT did not have any benefit, the trial is restricted to mMGMT patients.The CeTeG trial randomizes in a 1:1 fashion newly diagnosed GBM patients (18-70 years) for either standard TMZ therapy (concomitant and 6 courses à 4 weeks of adjuvant TMZ therapy) or experimental CCNU/TMZ therapy (6 courses à 6 weeks). Both arms include standard radiotherapy (RT) of the tumor site (30 x 2 Gy). Assuming that CCNU/TMZ therapy increases the median overall survival (mOS) from 48.9% (standard TMZ) to 70% (CCNU/TMZ; 75% in the previous phase II trial, Glas et al., 2009), 2 x 68 patients have to be accrued. Patients will be accrued over 24 months and each patient will be followed for at least 24 months adding up to a total minimal duration of the time from first patient in until the end of the follow-up time of 48 months. The primary endpoint is overall survival; secondary endpoints include progression-free survival, response rate, acute and late toxicity, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* patients have to be in a cognitive state that allows them to understand the rationale and necessity of study therapy and procedures.
* newly diagnosed histologically proven GBM or gliosarcoma WHO Grad IV
* methylated MGMT promoter in the tumor
* estimated life expectancy of at least 12 weeks
* Karnofsky Performance Score (KPS) ≥ 70%
* patient compliance and geographic proximity that allow adequate follow up
* male and female patients with reproductive potential must use an approved contraceptive method
* pre-menopausal female patients with childbearing potential: a negative serum pregnancy test must be obtained prior to treatment start
* Adequate organ function as described below:

Adequate bone marrow reserve:

white blood cell (WBC) count > 3000/µl, granulocyte count >1500/µl, platelets > 100000/µl, haemoglobin ≥ 10 g/dl Adequate liver function bilirubin < 1.5 times above upper limit of normal range (ULN), ALT and AST < 3 times ULN creatinine < 1.5 times ULN

Adequate blood clotting:

PT and PTT within normal limits Negative HIV test

Exclusion Criteria:

* prior malignancy
* prior chemotherapy
* prior radiotherapy to the brain
* concurrent administration of any other anti-tumor therapy
* allergy or other intolerability of temozolomide, CCNU, dacarbazine or other nitrosourea derivatives
* unable to undergo MRI
* past medical history of diseases with poor prognosis
* known HIV infection, active Hepatitis B or C infection
* any active infection
* female patients that are pregnant or breastfeeding
* patients with reproductive potential who do not accept to use contraception
* treatment in another clinical trial
* any psychological, cognitive, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up scheduled visits (at the discretion of investigator)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2010-10; Primary Completion 2017-04-06 (Actual); Study Completion 2017-04-06 (Actual)

PRIMARY OUTCOMES:
overall survival | after follow up (4 years)

SECONDARY OUTCOMES:
progression free survival | after follow up (4 years)
best response rate determined by MRI | after follow up (4 years)
frequency of delay of the next Lomustine/Temozolomide or Temozolomide course | during treatment period (2 years)
acute toxicity during radiotherapy and chemotherapy according to CTC AE V3.0 | during treatment period (2 years)
quality of life | including follow up (4 years)
Evaluation of late neurotoxicity | after follow up (4 years)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Herrlinger, Prof. Dr., Study Director — Division of Neurooncology, Departement of Neurology, University Hospital Bonn
Locations (12):
- Germany (12):
  - Depatment of Neurosurgery, Charité, University Hospital Berlin, Berlin
  - Department of Neurology, University Hospital Bochum, Bochum
  - Department of Neurology, University Hospital Bonn, Bonn
  - Department of Neurosurgery, University Hospital Cologne, Cologne
  - Department of Neurosurgery, University Hospital Dresden, Dresden
  - Department of Neurosurgery, University Hospital Duesseldorf, Düsseldorf
  - Department of Neurosurgery, University Hospital Frankfurt, Frankfurt
  - Department of Radiooncology, University Hospital Leipzig, Leipzig
  - Department of Neurosurgery, University of Heidelberg, Medical Faculty of Mannheim, Mannheim
  - Department of Neurosurgery, University Hospital Munich (LMU), Munich
  - Department of Neurosurgery, University Hospital Muenster, Münster
  - Department of Neurology, University Hospital Regensburg, Regensburg

REFERENCES:
- [Derived] Weller J, Schafer N, Schaub C, Tzaridis T, Zeyen T, Schneider M, Potthoff AL, Giordano FA, Steinbach JP, Zeiner PS, Kowalski T, Sabel M, Hau P, Krex D, Grauer O, Goldbrunner R, Schnell O, Tabatabai G, Ringel F, Schmidt-Graf F, Brehmer S, Tonn JC, Bullinger L, Vajkoczy P, Glas M, Vatter H, Herrlinger U, Seidel C. Patterns, predictors and prognostic relevance of high-grade hematotoxicity after temozolomide or temozolomide-lomustine in the CeTeG/NOA-09 trial. J Neurooncol. 2023 Jan;161(1):147-153. doi: 10.1007/s11060-022-04203-4. Epub 2023 Jan 7. PMID 36609807
- [Derived] Tzaridis T, Schafer N, Weller J, Steinbach JP, Schlegel U, Seidel S, Sabel M, Hau P, Seidel C, Krex D, Goldbrunner R, Tonn JC, Grauer O, Kebir S, Schneider M, Schaub C, Vatter H, Coch C, Glas M, Fimmers R, Pietsch T, Reifenberger G, Herrlinger U, Felsberg J. MGMT promoter methylation analysis for allocating combined CCNU/TMZ chemotherapy: Lessons learned from the CeTeG/NOA-09 trial. Int J Cancer. 2021 Apr 1;148(7):1695-1707. doi: 10.1002/ijc.33363. Epub 2020 Nov 10. PMID 33113214
- [Derived] Weller J, Tzaridis T, Mack F, Steinbach JP, Schlegel U, Hau P, Krex D, Grauer O, Goldbrunner R, Bahr O, Uhl M, Seidel C, Tabatabai G, Brehmer S, Bullinger L, Galldiks N, Schaub C, Kebir S, Stummer W, Simon M, Fimmers R, Coch C, Glas M, Herrlinger U, Schafer N. Health-related quality of life and neurocognitive functioning with lomustine-temozolomide versus temozolomide in patients with newly diagnosed, MGMT-methylated glioblastoma (CeTeG/NOA-09): a randomised, multicentre, open-label, phase 3 trial. Lancet Oncol. 2019 Oct;20(10):1444-1453. doi: 10.1016/S1470-2045(19)30502-9. Epub 2019 Sep 2. PMID 31488360
- [Derived] Herrlinger U, Tzaridis T, Mack F, Steinbach JP, Schlegel U, Sabel M, Hau P, Kortmann RD, Krex D, Grauer O, Goldbrunner R, Schnell O, Bahr O, Uhl M, Seidel C, Tabatabai G, Kowalski T, Ringel F, Schmidt-Graf F, Suchorska B, Brehmer S, Weyerbrock A, Renovanz M, Bullinger L, Galldiks N, Vajkoczy P, Misch M, Vatter H, Stuplich M, Schafer N, Kebir S, Weller J, Schaub C, Stummer W, Tonn JC, Simon M, Keil VC, Nelles M, Urbach H, Coenen M, Wick W, Weller M, Fimmers R, Schmid M, Hattingen E, Pietsch T, Coch C, Glas M; Neurooncology Working Group of the German Cancer Society. Lomustine-temozolomide combination therapy versus standard temozolomide therapy in patients with newly diagnosed glioblastoma with methylated MGMT promoter (CeTeG/NOA-09): a randomised, open-label, phase 3 trial. Lancet. 2019 Feb 16;393(10172):678-688. doi: 10.1016/S0140-6736(18)31791-4. Epub 2019 Feb 14. PMID 30782343
- See also: Clinical Neuro-Oncology, University of Bonn — http://neurologie.uni-bonn.de/forschungsbereiche/clinical-neurooncology.htm